CLINICAL TRIAL: NCT00577850
Title: Study to Determine the Pharmacokinetics of a Single 14C-labeled Intravenous Dose of Risedronate or Alendronate Followed by Once-a-week Unlabeled Oral Dose to Postmenopausal Women With Osteopenia or Osteoporosis
Brief Title: Pharmacokinetics of a Single 14C-labeled Dose of Risedronate or Alendronate Followed by Once-a-week Unlabeled Oral Dose
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Warner Chilcott (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2002095
Record Dates: First submitted 2007-12-19; First posted 2007-12-20 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Osteopenia; Osteoporosis
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis | interventions — Risedronic Acid; Alendronate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 0.23 mg 14C-labeled risedronate, followed 7 days later with oral 35 mg risedronate once a week for 52 weeks
  Interventions: Drug: risedronate
- 2 (Active Comparator): 0.45 mg 14C-labeled alendronate, followed 7 days later with oral 70 mg of alendronate once a week for 52 weeks
  Interventions: Drug: alendronate

INTERVENTIONS:
Drug: risedronate — 0.23 mg 14C-labeled risedronate, followed 7 days later with oral 35 mg risedronate once a week for 52 weeks followed by another 14C-labeled risedronate followed weekly by 35 mg risedronate for 3 weeks
  Arms: 1
Drug: alendronate — 0.45 mg 14C-labeled alendronate, followed 7 days later with oral 705 mg alendronate once a week for 52 weeks followed by another 14C-labeled alendronate followed weekly by 70 mg alendronate for 3 weeks
  Arms: 2

SUMMARY:
The primary objective of this study is to compare the urinary excretion of 14C-labeled risedronate and alendronate over 28 days.

ELIGIBILITY:
Inclusion Criteria:

* have medical history documentation verifying postmenopausal status of at least 2 years (natural or surgical). If not documented, confirmation will be required using estradiol < 20 pg/mL and follicle stimulating hormone (FSH) > 40 IU/mL;
* have osteopenia or osteoporosis (< 1.002 g/cm2 Lunar or < 0.882 g/cm2 Hologic) as determined by DXA of the lumbar spine (AP or PA view, L1-L4). This corresponds to a T-score of approximately < -1.5.

Exclusion Criteria:

* any clinically significant out-of-range laboratory values and vital signs,
* a clinically significant cardiovascular, hepatic, renal, or parathyroid disease, in the opinion of the Investigator
* a known hypersensitivity to bisphosphonates

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2002-11; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
compare the urinary excretion of 14C-labeled risedronate and alendronate over 28 days. | 28 days

SECONDARY OUTCOMES:
to compare urinary excretion and serum concentration-time profiles of 14C-labeled risedronate and alendronate over 52 weeks. | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Amy Sun, MD, PhD, Study Director — Procter and Gamble
Locations (2):
- United States (2):
  - Research Facility, Gainesville, Florida
  - Research Site, New Orleans, Louisiana